CLINICAL TRIAL: NCT04607356
Title: Blood Flow Restriction Exercise in the Treatment of Lateral Epicondylalgia vs Traditional Treatment
Brief Title: Blood Flow Restriction Exercise in the Treatment of Lateral Epicondylalgia Traditional Treatment
Acronym: BFR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tara Haugen, OTR/L, CBIS, LT, Physical Therapist, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NavalMCSD
Record Dates: First submitted 2020-10-13; First posted 2020-10-29 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Tennis Elbow; Lateral Epicondylitis
Keywords: Physical Therapy; Blood Flow Restriction; Tennis Elbow; Lateral Epicondylalgia
MeSH Terms: conditions — Tennis Elbow | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Outcomes Assessor
Masking Description: Treating therapists and patient will be aware of treatment. Grip strength objective measure will be performed by a clinician blinded to the participant's treatment group. All other outcome measures are patient-reported on outcome forms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Evidence-informed care (Active Comparator): Standardized, evidence based rehabilitation program for lateral epicondylalgia to include: discussion of ergonomics, home exercise program performance, use of any prescribed splint or brace, forearm and shoulder stretches, soft tissue mobilization, and performance of standard resistance exercises.
  Interventions: Other: Evidence-informed care
- Evidence-informed care + Blood Flow Restriction (BFR) (Experimental): Standardized, evidence based rehabilitation program for lateral epicondylalgia to include: discussion of ergonomics, home exercise program performance, use of any prescribed splint or brace, forearm and shoulder stretches, soft tissue mobilization, and performance of standard resistance exercises with the addition of BFR while performing resistive exercises.
  Interventions: Device: Blood Flow Restriction (BFR)

INTERVENTIONS:
Device: Blood Flow Restriction (BFR) — The Delphi Personalized Tourniquet System (PTS) will be utilized for the BFR exercises. The external constriction device will be applied to the proximal aspect of an individual's limb to restrict the flow of blood into and out of the extremity at 50% of usual flow. Subjects will perform a 30-15-15-15 repetition progression of 1-3 exercises as selected by the therapist. The Delphi PTS cuff is inflated at the start of the exercise and remains inflated throughout the exercise. Once the participant has completed an exercise, the cuff is deflated for 1 minute and the same cycle is performed for each subsequent exercise.
  Arms: Evidence-informed care + Blood Flow Restriction (BFR)
Other: Evidence-informed care — Evidence-based resistive exercises, stretches, soft tissue mobilization and patient education for lateral epicondylalgia.
  Arms: Evidence-informed care

SUMMARY:
The purpose of this study is to compare the clinical effectiveness and outcomes between current evidence based clinical care and use of personalized blood flow restriction training in the treatment of lateral epicondylalgia ("tennis elbow").

DETAILED DESCRIPTION:
Background: Lateral Epicondylalgia, or "tennis elbow", has been shown to affect up to 3% of the population and is a common musculoskeletal condition which also affects military service members. This study will compare clinical effectiveness of two treatment programs in individuals with lateral elbow pain.

Design: Prospective randomized controlled clinical trial

Methods: Participants, between the ages of 18-65, presenting to the NMCSD or NHCP Occupational or Physical Therapy Clinics with complaint of lateral elbow pain will be eligible for consideration to participate in this research. Patients that meet the inclusion criteria and elect to participate in the study will be randomized to either (1) a standardized, evidence based rehabilitation program or (2) an exercise volume matched group using personalized blood flow restriction (BFR) exercise.

Upon entry to the program subjects will complete measurements of height, body weight, physical activity level (Marx Activity Scale), annotation of their dominant upper extremity (UE), the patient-rated tennis elbow evaluation (PRTEE) questionnaire, Numerical Pain Rating Scale (NPRS), Patient-Reported Outcome Measurement Information System version 1.2- Global Health (PROMIS scale v1.2- Global Health), and grip strength using the JAMAR dynamometer. At the end of each treatment session subjects will complete the Numerical Pain Rating Scale (NPRS) and the OMNI-Resistance Exercise Scale (OMNI-RES) rating of perceived exertion (RPE) survey.

The standard rehabilitation group will perform active wrist extension, forearm supination, and gripping. These exercises may include isometric, concentric, or eccentric forms of strengthening contingent upon clinical decision making. Specifics of exercise performance (to include magnitude of resistance and volume of exercise) will be documented in the treatment record.

The Delphi Personalized Tourniquet System (PTS) will be utilized for the BFR exercises. The Delphi PTS measures an individual's personalized tourniquet pressure (PTP) using doppler technology similar to a blood pressure cuff. In the BFR exercise condition, subjects will perform a 30-15-15-15 repetition progression of 1-3 exercises as selected by the therapist.

Participants will be provided in-clinic treatment for a maximum of 12 sessions, one to three treatment sessions weekly, and may be discharged prior to that based upon shared decision making between the participant and therapist. The NPRS, grip strength, PROMIS scale v1.2- Global Health, and PRTEE will be completed at the last clinical appointment, as well as three and six-week, and three and six month follow up appointments. Twelve months following completion of occupational/physical therapy clinical care participants will be contacted and asked to complete a verbal NPRS, PROMIS scale v1.2- Global Health and the PRTEE outcome scale. Additionally, at 12 months following discharge from Physical or Occupational Therapy, the participants' EMR will be reviewed for follow-up visits related to the same condition (LET).

Data Analysis: A mixed effects longitudinal model will be utilized to assess for differences in the primary outcome measures (grip strength, NPRS, and PRTEE) between the time points of intake, end of occupational/physical therapy treatment, and three and six months post completion of treatment. Secondary analysis of change in OMNI-RES RPE and NPRS during the course of treatment will also be analyzed with a mixed effects longitudinal model. Healthcare provider(s) will be analyzed as a co-variate. Microsoft Excel and SPSS will function as the main data analysis instruments.

Clinical Implications: Results of this study are expected to guide clinician's selection of rehabilitation techniques to improve outcomes (increase strength, improve function, and decrease pain), improve mission readiness by earlier return to duty, reduce healthcare service costs, and also reduce lost duty/work time.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of lateral elbow pain (e.g. "tennis elbow" or wrist extensor tendinopathy)
2. Between the ages of 18-65
3. Elbow pain for 4 weeks or more

Exclusion Criteria:

1. Ligamentous elbow sprain, osteoarthritis of elbow and cervical radiculopathy in the affected limb will be excluded from the study.
2. Any history of ligamentous, bony or other soft tissue reconstruction surgery at the affected elbow.
3. Vascular disorders to include: history of DVT, history of endothelial dysfunction, peripheral vascular disease
4. Current fracture in affected arm
5. History of crush injury to affected arm
6. Any surgery on affected arm in last 1 year
7. Surgery within last year on contralateral upper extremity
8. History of lymphectomy (such as axillary exploration with breast surgery, lymph node biopsy in the affected axilla/arm)
9. Pregnancy
10. Active infection
11. Current cancer diagnosis/treatment
12. Sickle cell anemia or trait
13. Kidney dialysis
14. History of syncope/passing out with pressure to body (such as massage, or blood pressure cuff).
15. Inability to consent
16. Thromboembolism
17. Varicose veins
18. Cardiovascular disorders
19. Taking anti-coagulant medications
20. Bleeding disorder
21. Instructed by a physician or medical practitioner that they are not cleared to exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | Taken at initial intake, after completion of each treatment session (up to 12 total sessions following initial evaluation), and at the 3-week, 6-week, 3-month, 6-month and 12-month followup sessions
  Change in score on 0-10 pain rating scale with 0 being no pain, and 10 being worst pain
Patient-rated tennis elbow evaluation (PRTEE) | Taken at initial intake, and at the 3-week, 6-week, 3-month, 6-month and 12-month followup sessions
  Change in score of the patient reported outcome measure (form): rating pain as well as difficulty on a scale of 0-10 with certain movements and functional activities. Lower numbers suggest less pain, higher scores suggest more pain. Total score 0-100.
Grip Strength | Taken at initial intake, and at the 3-week, 6-week, 3-month, and 6-month follow-up sessions
  Assessing change in grip strength using the JAMAR dynamometer- taken with elbow straight, average of 3 measurements recorded.

SECONDARY OUTCOMES:
Patient-Reported Outcome Measurement Information System version 1.2- Global Health | Taken at initial intake, and at the 3-week, 6-week, 3-month, 6-month and 12-month followup sessions
  Looking at mental health factors

CONTACTS AND LOCATIONS:
Overall Officials: Tara Haugen, MSOT, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Navy Medical Readiness & Training Command San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Result] Loenneke JP, Wilson JM, Wilson GJ, Pujol TJ, Bemben MG. Potential safety issues with blood flow restriction training. Scand J Med Sci Sports. 2011 Aug;21(4):510-8. doi: 10.1111/j.1600-0838.2010.01290.x. Epub 2011 Mar 16. PMID 21410544
- [Result] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Result] Slysz J, Stultz J, Burr JF. The efficacy of blood flow restricted exercise: A systematic review & meta-analysis. J Sci Med Sport. 2016 Aug;19(8):669-75. doi: 10.1016/j.jsams.2015.09.005. Epub 2015 Sep 28. PMID 26463594
- [Result] Yasuda T, Brechue WF, Fujita T, Shirakawa J, Sato Y, Abe T. Muscle activation during low-intensity muscle contractions with restricted blood flow. J Sports Sci. 2009 Mar;27(5):479-89. doi: 10.1080/02640410802626567. PMID 19253083
- [Result] Day JM, Lucado AM, Uhl TL. A COMPREHENSIVE REHABILITATION PROGRAM FOR TREATING LATERAL ELBOW TENDINOPATHY. Int J Sports Phys Ther. 2019 Sep;14(5):818-829. PMID 31598419